CLINICAL TRIAL: NCT04881721
Title: Mesh-free Suture Urethropexy for Treating Stress Urinary Incontinence, Efficacy and Durability Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Ghazaleh Rostami Nia, Director of Research Division of Urogynecology, NorthShore University HealthSystem, Endeavor Health
Other Study IDs: EH21-062
Record Dates: First submitted 2021-04-08; First posted 2021-05-11 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Urethropexy — Suture based (Mesh-free) surgery to stabilize the urethra for the treatment of stress urinary incontinence

SUMMARY:
In this proposed study, the investigators aim to evaluate a modified suture urethropexy technique for the treatment of female stress urinary incontinence.

Participants will be followed with postoperative visits after 2 weeks, 2 months, and 12 months. Pelvic floor ultrasound imaging will be performed before surgery and after 2 months and 12 months, to evaluate urethral mobility.

DETAILED DESCRIPTION:
This study is designed as a prospective observational study. The hypothesis is that suture urethropexy will improve stress urinary incontinence symptoms in participants with stress urinary incontinence and normal urethral closure pressure at 2 months and 12 months after surgery.

Specific Aims:

Aim 1: Investigate the efficacy of this mesh-free suture based surgical technique for improving SUI symptoms

Aim 2: Investigate the efficacy of this mesh-free suture based surgical technique on key urethral support defects observed with 3D ultrasound

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with stress dominant urinary incontinence
* Stress urinary incontinence confirmed by testing (e.g. urodynamics)
* Able to provide informed consent and attend post-operative visits

Exclusion Criteria:

* Detrusor overactivity (> 40cm H2O)
* Maximum Urethral Closure Pressure (< 40 cm H2O)
* Post void residual > 150 mL
* Prior surgery for stress urinary incontinence with retained material (e.g. bulking agent, sling)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with female pelvic anatomy, 18 years or older, with stress dominant urinary incontinence interested and eligible for surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress urinary incontinence symptoms | 2 weeks
  Severity of stress urinary incontinence symptoms by questionnaire
Stress urinary incontinence symptoms | 3 months
  Severity of stress urinary incontinence symptoms by questionnaire
Stress urinary incontinence symptoms | 12 months
  Severity of stress urinary incontinence symptoms by questionnaire
Voiding dysfunction | Within 1 year of surgery
  Rate of urinary retention after surgery

SECONDARY OUTCOMES:
Distal Urethral Motion | 2 months
  Distal urethral swing angle during Valsalva measured via pelvic ultrasound
Distal Urethral Motion | 12 months
  Distal urethral swing angle during Valsalva measured via pelvic ultrasound
Proximal Urethral Motion | 2 months
  Proximal urethral swing angle during Valsalva measured via pelvic ultrasound
Proximal Urethral Motion | 12 months
  Proximal urethral swing angle during Valsalva measured via pelvic ultrasound
Post-operative complications | Within 1 year of surgery
  Rate of post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Rostami Nia, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford AA, Rogerson L, Cody JD, Aluko P, Ogah JA. Mid-urethral sling operations for stress urinary incontinence in women. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD006375. doi: 10.1002/14651858.CD006375.pub4. PMID 28756647
- [Background] Richter HE, Albo ME, Zyczynski HM, Kenton K, Norton PA, Sirls LT, Kraus SR, Chai TC, Lemack GE, Dandreo KJ, Varner RE, Menefee S, Ghetti C, Brubaker L, Nygaard I, Khandwala S, Rozanski TA, Johnson H, Schaffer J, Stoddard AM, Holley RL, Nager CW, Moalli P, Mueller E, Arisco AM, Corton M, Tennstedt S, Chang TD, Gormley EA, Litman HJ; Urinary Incontinence Treatment Network. Retropubic versus transobturator midurethral slings for stress incontinence. N Engl J Med. 2010 Jun 3;362(22):2066-76. doi: 10.1056/NEJMoa0912658. Epub 2010 May 17. PMID 20479459
- [Background] Kenton K, Stoddard AM, Zyczynski H, Albo M, Rickey L, Norton P, Wai C, Kraus SR, Sirls LT, Kusek JW, Litman HJ, Chang RP, Richter HE. 5-year longitudinal followup after retropubic and transobturator mid urethral slings. J Urol. 2015 Jan;193(1):203-10. doi: 10.1016/j.juro.2014.08.089. Epub 2014 Aug 23. PMID 25158274
- [Background] Nolfi AL, Brown BN, Liang R, Palcsey SL, Bonidie MJ, Abramowitch SD, Moalli PA. Host response to synthetic mesh in women with mesh complications. Am J Obstet Gynecol. 2016 Aug;215(2):206.e1-8. doi: 10.1016/j.ajog.2016.04.008. Epub 2016 Apr 16. PMID 27094962
- [Background] Frenkl TL, Rackley RR, Vasavada SP, Goldman HB. Management of iatrogenic foreign bodies of the bladder and urethra following pelvic floor surgery. Neurourol Urodyn. 2008;27(6):491-5. doi: 10.1002/nau.20558. PMID 18537142
- [Background] Brubaker L, Norton PA, Albo ME, Chai TC, Dandreo KJ, Lloyd KL, Lowder JL, Sirls LT, Lemack GE, Arisco AM, Xu Y, Kusek JW; Urinary Incontinence Treatment Network. Adverse events over two years after retropubic or transobturator midurethral sling surgery: findings from the Trial of Midurethral Slings (TOMUS) study. Am J Obstet Gynecol. 2011 Nov;205(5):498.e1-6. doi: 10.1016/j.ajog.2011.07.011. Epub 2011 Jul 20. PMID 21925636
- [Background] Baracat F, Mitre AI, Kanashiro H, Montellato NI. Endoscopic treatment of vesical and urethral perforations after tension-free vaginal tape (TVT) procedure for female stress urinary incontinence. Clinics (Sao Paulo). 2005 Oct;60(5):397-400. doi: 10.1590/s1807-59322005000500008. Epub 2005 Oct 24. PMID 16254676
- [Background] Giri SK, Drumm J, Flood HD. Endoscopic holmium laser excision of intravesical tension-free vaginal tape and polypropylene suture after anti-incontinence procedures. J Urol. 2005 Oct;174(4 Pt 1):1306-7. doi: 10.1097/01.ju.0000173926.04596.55. PMID 16145408
- [Background] Koduri S, Goldberg RP, Sand PK. Transvaginal therapy of genuine stress incontinence. Urology. 2000 Dec 4;56(6 Suppl 1):23-7. doi: 10.1016/s0090-4295(00)00509-4. PMID 11114559